CLINICAL TRIAL: NCT06685926
Title: Groin-Only Lymphaticovenous Anastomosis for Lower Extremity Lymphoedema: a Retrospective Cohort Propensity-Score Matched Analysis of a Novel Supermicrosurgical Concept
Brief Title: The Impact of Supermicrosurgery Intervention on Patients with Lower Extremity Lymphedema Using Groin-Only Approach Lymphaticovenous Anastomosis
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202401630B0
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Lymphedema; Lymphedema of Leg
Keywords: propensity score matching; LVA; supermicrosurgery; lymphaticovenous anastomosis; lymphovenous bypass
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Groin-Only Approach LVA: This is a group of patients who had a single incision based LVA procedure.
  Interventions: Procedure: Supermicrosurgical LVA, Groin Approach Only (lymphatic vessel to recipient vien lumen-to-lumen anastomosis)
- Conventional Approach LVA: This is a group of patients who had the conventional LVA approach with multiple incisions for access.
  Interventions: Procedure: Supermicrosurgical LVA, Conventional Multiple Access Approach Only (lymphatic vessel to recipient vien lumen-to-lumen anastomosis)

INTERVENTIONS:
Procedure: Supermicrosurgical LVA, Groin Approach Only (lymphatic vessel to recipient vien lumen-to-lumen anastomosis)
  Groups: Groin-Only Approach LVA
Procedure: Supermicrosurgical LVA, Conventional Multiple Access Approach Only (lymphatic vessel to recipient vien lumen-to-lumen anastomosis)
  Groups: Conventional Approach LVA

SUMMARY:
This study employs a propensity score-matched analysis to compare the treatment outcomes, focusing on percentage volume reduction between the conventional multi-incision lymphaticovenous anastomosis (LVA) technique and the novel single groin incision LVA technique in patients with unilateral lower extremity lymphoedema.

DETAILED DESCRIPTION:
Lymphaticovenous anastomosis (LVA), a surgical technique that connects lymphatic vessels (LVs) to adjacent veins, has demonstrated efficacy in alleviating lymphedema by enabling the drainage of stagnant lymphatic fluid.

Conventional LVA treatment for lower extremity lymphoedema (LEL) has favored distal, multiple incisions in the lower leg due to the denser and more superficial distribution of LVs and recipient veins in the distal regions.

Based on the recent advancement in the understaning of lymphosomes and the role of antegrade lymph flow, a shift to more proximal LVA around the groin region for LEL could be theoretically advantagous, but its clinical efficacy compared to conventional distal LVA remains underexplored.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lymphatic-related diseases to the lower extremity
* Patients who is undergoing LVA for unilateral lower-limb lymphedema.

Exclusion Criteria:

* Primary lymphedema
* Bilateral lower limb lymphedema
* History of previous treatment for lymphedema (LVA, vascularized lymph node transfer (VLNT), liposuction, or excisional therapy such as the Charles procedure) - Those that were lost to follow-up.
* Patients who recieved both LVA to the groin site and non-groin site.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2024-09 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Volume change after LVA | 6 and 12 months
  The primary endpoint is limb volume change at 6 and 12 months after intervention, measured using magnetic resonance volumetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No